CLINICAL TRIAL: NCT00016367
Title: Phase II Multidose, Single Arm, Multicenter Clinical Trial of Cisplatin and Gemcitabine in Combination With Recombinant Humanized Anti-p185HER2 Monoclonal Antibody (Herceptin) in Patients Who Have Untreated p185HER2 Overexpressing Advanced Local Stage (Stage IIIb Pleural Effusion Only) and Metastatic (Stage IV) Non-Small Cell Lung Cancer
Brief Title: Cisplatin and Gemcitabine Plus Trastuzumab in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM99-015; P30CA016672 (NIH); MDA-DM-99015 (Other: UT MD Anderson Cancer Center); NCI-4450; CDR0000068626 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2001-05-06; First posted 2004-02-27 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Trastuzumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen A (Experimental): Gemcitabine IV followed by Cisplatin IV Day 1 and Trastuzumab (Herceptin) IV Day 2; Trastuzumab IV followed by Gemcitabine IV Day 8 and Trastuzumab IV Day 15.
  Interventions: Biological: Trastuzumab; Drug: Cisplatin; Drug: Gemcitabine Hydrochloride
- Regimen B (Experimental): Starting Day 22 of regimen A, Trastuzumab IV, Gemcitabine IV, and Cisplatin IV Day 1. Trastuzumab IV followed by Gemcitabine IV Day 8 and Trastuzumab IV Day 15. Repeats every 21 days for up to 5 courses.
  Interventions: Biological: Trastuzumab; Drug: Cisplatin; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Biological: Trastuzumab — Regimen A: Trastuzumab IV over 90 minutes on days 2 and 8.
  Regimen B: Trastuzumab IV over 30-90 minutes on days 1, 8 and 15.
  Other Names: Herceptin
Drug: Cisplatin — Regimen A: Cisplatin IV over 2 hours on day 1 following gemcitabine.
  Regimen B: Cisplatin IV over 2 hours on day 1.
  Other Names: Platinol; Platinol-AQ; CDDP
Drug: Gemcitabine Hydrochloride — Regimen A: Gemcitabine IV over 30 minutes on day 1. Gemcitabine IV over 30 minutes on day 8 following Trastuzumab.
  Regimen B: Gemcitabine IV over 30 minutes on day 1. Gemcitabine IV over 30 minutes on day 8 following Trastuzumab.
  Other Names: Gemzar; Gemcitabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining chemotherapy with monoclonal antibody therapy may kill more tumor cells.

PURPOSE: Phase II trial to study effectiveness of combining cisplatin, gemcitabine, and trastuzumab in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the therapeutic efficacy and toxicity of cisplatin, gemcitabine, and trastuzumab (Herceptin) in patients with untreated p185-HER2 overexpressing stage IIIB or IV non-small cell lung cancer. II. Determine the pharmacokinetic interactions among these drugs in these patients. III. Assess the pharmacodynamics of these drugs in these patients.

OUTLINE: This is a multicenter study. Regimen A: Patients receive gemcitabine IV over 30 minutes followed by cisplatin IV over 2 hours on day 1 and trastuzumab (Herceptin) IV over 90 minutes on day 2. Patients receive trastuzumab IV over 90 minutes followed by gemcitabine IV over 30 minutes on day 8 and trastuzumab IV over 90 minutes on day 15. Patients proceed to regimen B on day 22 of regimen A. Regimen B: Patients receive trastuzumab IV over 30-90 minutes, gemcitabine IV over 30 minutes, and cisplatin IV over 2 hours on day 1. Patients receive trastuzumab IV over 30-90 minutes followed by gemcitabine IV over 30 minutes on day 8 and trastuzumab IV over 30-90 minutes on day 15. Treatment repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity. Maintenance: After completion of 6 courses, patients with stable disease or partial response receive trastuzumab IV over 30-90 minutes weekly until tumor progression.

PROJECTED ACCRUAL: A total of 20-48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Immunohistochemically confirmed p185-HER2 expressing stage IIIB (pleural effusions only) or IV non-small cell lung cancer Confirmed overexpression at least: 1+ p185-HER2 (by DAKO Hercep Test) OR 15 ng/mL serum HER2/neu shed antigen (by Human HER2 Quantitative ELISA) At least 1 site of measurable disease outside of prior radiation port Brain metastases allowed provided clinical neurologic status is stable and head CT scan is stable to improved

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Zubrod 0-2 Life expectancy: More than 12 weeks Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL (transfusion allowed) Hepatic: Bilirubin less than 1.5 mg/dL SGPT no greater than 1.5 times normal Renal: Creatinine clearance at least 60 mL/min Cardiovascular: No myocardial infarction within the past 6 months No unstable angina, uncontrolled congestive heart failure, or uncontrolled arrhythmia Ejection fraction at least 40% Other: No other malignancy within the past 5 years No concurrent serious infection, including post-obstructive pneumonia No more than 10% weight loss in past 3 months Not pregnant or nursing Negative pregnancy test Fertile patients must use adequate contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 3 weeks since prior radiotherapy (including radiotherapy for brain metastases) No concurrent radiotherapy to only site of measurable disease Surgery: At least 2 weeks since prior major surgery No concurrent surgery on only site of measurable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 1999-05-13 (Actual); Primary Completion 2004-12-14 (Actual); Study Completion 2004-12-14 (Actual)

PRIMARY OUTCOMES:
Efficacy of Cisplatin, Gemcitabine, + Trastuzumab in Untreated p185-HER2 Overexpressing Stage IIIB or IV Non-small Cell Lung Cancer | 21 days cycles for 6 courses

CONTACTS AND LOCATIONS:
Overall Officials: Roy S. Herbst, MD, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org